CLINICAL TRIAL: NCT00852592
Title: Efficacy of Light Therapy for Bipolar Depression: A Randomized Controlled Trial
Brief Title: Light Therapy for Bipolar Disorder. Efficacy of Light Therapy for Bipolar Depression: A Randomized Controlled Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Dorothy Sit, Associate Professor of Psychiatry and Behavioral Sciences, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO09020546
Record Dates: First submitted 2009-02-25; First posted 2009-02-27 (Estimated); Results first posted 2016-11-07 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-09

CONDITIONS: Bipolar Disorder; Major Depressive Episode
Keywords: Bipolar Disorder Depression Midday Light Therapy; Bipolar Disorder Type I or II
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Comparator (Active Comparator): 7000lux broad-spectrum light
  Interventions: Device: 7000lux broad-spectrum light
- Inactive Comparator (Placebo Comparator): 50lux dim red light
  Interventions: Device: 50lux dim red light

INTERVENTIONS:
Device: 7000lux broad-spectrum light — dosage - 15-60minutes NOON-2PM daily
  Arms: Active Comparator
Device: 50lux dim red light — dosage: 15-60minutes NOON-2PM daily
  Arms: Inactive Comparator

SUMMARY:
The purpose of this study is to understand the efficacy of light therapy for bipolar depression.

DETAILED DESCRIPTION:
Bipolar Disorders (BD) are associated with chronic depression, disability, and increased suicide risk. Building on earlier findings, we conducted a 6-week randomized, double-blind, placebo-controlled trial to investigate the efficacy of midday light therapy for bipolar depression. The aims were to examine the change in depression levels and the proportion of patients who responded and remitted. We assessed predictors of response with measures of side effects, sleep quality, suicidality, and psychosocial functioning. We included depressed adults with BD-Type I or II confirmed on the SCID interview and taking stable-dosed antimanic medication. We excluded patients with psychosis, rapid cycling, obsessive compulsive disorder, alcohol or substance use disorders, hypomania or mania, and severe suicidality. Patients were randomized to 7000 lux broad spectrum light therapy OR 50 lux dim red light for 45-60 minutes daily. Weekly, the blinded-clinician assessed symptoms with the Structured Interview Guide for the Hamilton Depression Scale with Atypical Depression Supplement (SIGH-ADS) and global functioning.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65 years
* DSM-IV Criteria BD I or II depressive episode,
* SIGH-ADS >20; duration >2 weeks.
* Stable dose antidepressant drug >8 weeks with concurrent antimanic drug
* Controlled thyroid disease
* Subjects with preexisting eye diseases will be included.
* Able to provide informed consent
* Stable minimum dose antimanic drug >4weeks: lithium 0.5 mEq/L, divalproex Na 50 mcg/mL, olanzapine 5mg daily, carbamazepine 4mg/L; lamotrigine 100mg daily, risperidone 2mg daily, quetiapine 400 mg daily, ziprasidone 10 mg bid, and aripiprazole 5 mg qd.
* Stable unchanged psychotherapy for >16weeks

Exclusion Criteria:

* The following eye diseases: retinal disease, cataract surgery and lens removal, macular degeneration,
* Taking photosensitizing drugs such as phenothiazines (chlorpromazine), antimalarial drugs, melatonin and hypericum.
* Acute psychosis (DSM-IV Criteria)
* Rapid cycling in the past 1 year
* Obsessive compulsive disorder
* Alcohol or substance abuse or dependence in the past 6 months.
* MRS>5
* Recent history of a suicide attempt (3 months) or active suicidal Ideation (SIGHADS item H11 >2)
* Beta-adrenergic blockers, exogenous melatonin, chronic NSAIDS

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-05; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy K Sit, M.D., Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - University of Pittsburgh, Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided
We can share data if approached by other investigators

REFERENCES:
- [Derived] Sit DK, McGowan J, Wiltrout C, Diler RS, Dills JJ, Luther J, Yang A, Ciolino JD, Seltman H, Wisniewski SR, Terman M, Wisner KL. Adjunctive Bright Light Therapy for Bipolar Depression: A Randomized Double-Blind Placebo-Controlled Trial. Am J Psychiatry. 2018 Feb 1;175(2):131-139. doi: 10.1176/appi.ajp.2017.16101200. Epub 2017 Oct 3. PMID 28969438

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Light Unit: active light therapy unit: dosage - 15-60minutes NOON-2PM daily
- Inactive Light Unit: Inactive light therapy unit: dosage: 15-60minutes NOON-2PM daily
Period: Overall Study
Arm/Group | Active Light Unit | Inactive Light Unit
Started | 23 | 23
Completed | 20 | 19
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Active Comparator: active light unit
  active light therapy unit: dosage - 15-60minutes NOON-2PM daily
- Inactive Comparator: inactive light unit
  Inactive light therapy unit: dosage: 15-60minutes NOON-2PM daily
- Total: Total of all reporting groups
Arm/Group | Active Comparator | Inactive Comparator | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 23 | 46
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (12) | 45 (15) | 44 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 8 | 7 | 15
Region of Enrollment [Number; unit: participants]
  United States | 23 | 23 | 46
SIGH-ADS depression score [Mean (Standard Deviation); unit: units on a scale] — The Structured Interview Guide for the Hamilton Depression Rating Scale-HRS-D with Atypical Depression Supplement (SIGH-ADS) provides a benchmark for depression severity; SIGH-ADS scores range from 0-79; higher values represent increased depression severity and worse outcome.
  units on a scale | 26.1 (5.2) | 30.1 (6.1) | 28.1 (5.9)
Global Assessment of Functioning (GAF) [Mean (Standard Deviation); unit: units on a scale] — The Global Assessment of Function (GAF) was used to assess psychosocial functioning. Scores range from 0-100 with higher values representing higher functioning and better outcome.
  units on a scale | 57.4 (5.61) | 53.5 (5.32) | 55.4 (5.76)

OUTCOME MEASURES:

1. Primary Outcome: SIGH-ADS Depression Score
Description: The Structured Interview Guide for the Hamilton Depression Rating Scale-HRS-D with Atypical Depression Supplement (SIGH-ADS) provides a benchmark for depression severity; SIGH-ADS scores range from 0-79; higher values represent increased depression severity and worse outcome.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Light Unit | Inactive Light Unit
Number analyzed (Participants) | 23 | 23
units on a scale | 10.3 (8.18) | 17.3 (9.53)
Statistical Analysis 1: Comparison: Active Light Unit vs Inactive Light Unit; Test type: Superiority or Other; p = 0.005, ANOVA

2. Secondary Outcome: Global Assessment of Functioning (GAF)
Description: The GAF is used to assess global psychosocial functioning. Scores range from 0-100 with higher values representing higher functioning and better outcome.
Time Frame: 6-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Light Unit | Inactive Light Unit
Number analyzed (Participants) | 23 | 23
units on a scale | 73.9 (9.77) | 65.2 (9.83)
Statistical Analysis 1: Comparison: Active Light Unit vs Inactive Light Unit; Test type: Superiority or Other; p = 0.004, ANOVA

ADVERSE EVENTS:
Arm/Group | Active Comparator | Inactive Comparator
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes